CLINICAL TRIAL: NCT01801982
Title: A Follow Up Investigation For Patients Completing Study A1481276 To Investigate Developmental Progress 12 And 24 Months Following Completion Of Sildenafil Treatment
Brief Title: A Non-Interventional Follow Up Study For Subjects Who Received Sildenafil for Persistent Pulmonary Hypertension of the Newborn (PPHN)
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481283; 2010-021266-30 (EudraCT Number)
Record Dates: First submitted 2013-01-08; First posted 2013-03-01 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Hypertension, Persistent, of the Newborn
Keywords: PPHN; development progress after PPHN; developmental progress after sildenafil.
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: non-interventional — non-interventional

SUMMARY:
This single center study will monitor the developmental progress of PPHN patients who received iv sildenafil in study A1481276. Two visits will be conducted, at 12 and 24 months following the end of study drug infusion.

DETAILED DESCRIPTION:
This study will monitor developmental progress of PPHN patients for 2 years following study treatment, using Bayley III and Hammersmith tools. Data will be explored with descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Any subject who received sildenafil treatment in study A1481276.
* Signed and dated informed consent document by legal guardian.

Exclusion Criteria:

* Any subject who did not receive sildenafil treatment during study A1481276.

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients who took part in study A1481276 following PPHN treatment with IV sildenafil
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Great Ormond Street Hospital, Paediatric Intensive Care, London, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481283&StudyName=A%20Non-Interventional%20Follow%20Up%20Study%20For%20Subjects%20Who%20Received%20Sildenafil%20for%20Persistent%20Pulmonary%20Hypertension%20of%20the%20Newborn%20%28PPHN%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants who received sildenafil treatment during study A1481276 (NCT01069861) were eligible for enrollment in this study.
Groups:
- Sildenafil: Participants who received intravenous (IV) sildenafil treatment in study A1481276 (NCT01069861) were followed-up for safety, up to Month 24.
Period: Overall Study
Arm/Group | Sildenafil
Started | 1
Completed | 0
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all enrolled participants.
Arm/Group | Sildenafil
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.2 (NA) — Standard Deviation was not reported as only 1 participant was evaluated.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Physical Examination Abnormalities at Month 12
Description: Physical examinations included height, weight, head circumference, general appearance, skin examination, abdominal examination, respiratory system, neurological examination, hearing and ophthalmology assessments. Physical examination abnormalities were based on investigator discretion.
Time Frame: Month 12
Population: Full Analysis Set (FAS) included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 1
participants | 0

2. Primary Outcome: Number of Participants With Physical Examination Abnormalities at Month 24
Description: as for outcome 1
Time Frame: Month 24
Population: Data was not possible to report as participant lost to follow-up at Month 24 (Visit 2) after Month 12 follow-up (Visit 1).
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants With Clinically Significant Medical History at Month 12
Description: Criteria for clinically significant medical history included any hospital admissions or any medications given since discharge from Study A1481276 (NCT01069861) that were considered clinically significant by the investigator.
Time Frame: Month 12
Population: Full Analysis Set (FAS) included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 1
participants | 0

4. Primary Outcome: Number of Participants With Clinically Significant Medical History at Month 24
Description: as for outcome 3
Time Frame: Month 24
Population: as for outcome 2
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival at Month 12
Description: Overall survival was the duration from enrollment to death. For participants who are alive, overall survival was censored at the last contact. Number of participants who were alive at Month 12 was to be reported.
Time Frame: Month 12
Population: Full Analysis Set (FAS) included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 1
participants | 1

6. Secondary Outcome: Overall Survival at Month 24
Description: Overall survival was the duration from enrollment to death. For participants who are alive, overall survival was censored at the last contact. Number of participants who were alive at Month 24 was to be reported.
Time Frame: Month 24
Population: as for outcome 2
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to Month 12
Population: FAS included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Sildenafil
Number analyzed (Participants) | 1
participants | 0

ADVERSE EVENTS:
Arm/Group | Sildenafil
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Results at Month 24 were not reported as the participant lost to follow-up after Month 12.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.